CLINICAL TRIAL: NCT03685357
Title: Investigation of the Possible Correlation Between Idiopathic Parkinson's Disease and Diabetes Mellitus in Egyptian Elderly Patients
Brief Title: Correlation Between Idiopathic Parkinson's Disease and Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Collaborators: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Afnan Awad-Allah Elgnainy, Master student, teaching assistant of Clinical Pharmacy, Ain Shams University
Other Study IDs: AinShamsUni Afnan
Record Dates: First submitted 2018-09-22; First posted 2018-09-26 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood Samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Idiopathic Parkinson's: Oral glucose tolerance test
  The Unified Parkinson's Disease Rating Scale (UDPRS).
- Diabetics receive sulphonylurea group: Record RBDSQ ("Rapid eye movement Sleep" Behavior Disorder Screening Questionnaire) total score
- Diabetics on sulphonylurea and metformin: Record RBDSQ ("Rapid eye movement Sleep" Behavior Disorder Screening Questionnaire) total score
- Healthy: Record RBDSQ ("Rapid eye movement Sleep" Behavior Disorder Screening Questionnaire) total score
  Oral glucose tolerance test

SUMMARY:
Correlation between Idiopathic Parkinson's disease and diabetes mellitus in Egyptian Elderly Patients

DETAILED DESCRIPTION:
1. Record RBDSQ ("Rapid eye movement Sleep" Behavior Disorder Screening Questionnaire) total score difference between Group 1 and Group 2 .
2. Oral glucose tolerance test will be performed and compared between Group 3 and Group 4.
3. Association between glucose level and motor complication of L-dopa among Idiopathic Parkinson's patients using Unified Parkinson's Disease Rating Scale (UDPRS).

ELIGIBILITY:
Inclusion Criteria:

1. Diabetic Patients
2. Idiopathic Parkinsonism

Exclusion Criteria:

1. Secondary Parkinsonism due to stroke, trauma and encephalitis.
2. Drug induced Parkinsonism.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Egyptian Elderly
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
UPDRS (Unified Parkinson's Disease Rating) Scale) | Baseline
  Association between glucose level and motor complication of L-dopa among Idiopathic , , Parkinson's patients using Unified Parkinson's Disease Rating Scale (UDPRS)., high scores mean worsen condition
Oral Glucose Tolerance Test | 0, 0.5 hour , 1 hour, 1.5 hour , 2 hour
  Between Idiopathic Parkinson's patients and the Control group
RBDSQ ("Rapid eye movement Sleep" Behavior Disorder Screening Questionnaire) | Baseline
  among Diabetic Patients, total score 13 , high scores mean worsen condition

CONTACTS AND LOCATIONS:
Overall Officials: Afnan Elgnainy, Principal Investigator — AinShams University
Locations (1):
- AinShams University, Cairo, Egypt

REFERENCES:
- [Derived] AwadAllah Elgnainy A, Hamed MI, Osman Mohamed W, Sabri NA. Investigation of the Possible Correlation between Idiopathic Parkinson's Disease and Diabetes Mellitus in Egyptian Patients: A Pilot Study. Neurol Res Int. 2021 Nov 12;2021:2838669. doi: 10.1155/2021/2838669. eCollection 2021. PMID 34804608